CLINICAL TRIAL: NCT05762237
Title: Prediction of Intraoperative Hypotension Using Non-invasive Monitoring Devices: Development of Deep Learning Model
Brief Title: Deep Learning Models for Prediction of Intraoperative Hypotension Using Non-invasive Parameters
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Professor, Samsung Medical Center
Other Study IDs: SMC 2022-09-096
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Intraoperative Hypotension; General Anesthesia
Keywords: intraoperative hypotension; noninvasive monitor; deep learning algorithm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: In the open source database (VitalDB, https://vitaldb.net), the patients who underwent general anesthesia with non-invasive monitoring including blood pressure, electrocardiography, pulse oximetry, bispectral index, capnography, and minimal alveolar concentration of inhalation agent.

SUMMARY:
The investigators aimed to investigate the deep learning model to predict intraoperative hypotension using non-invasive monitoring parameters.

DETAILED DESCRIPTION:
Intraoperative hypotension is associated with various postoperative complications such as acute kidney injury. Therefore, precise prediction and prompt treatment of intraoperative hypotension are important. However, it is difficult to accurately predict intraoperative hypotension based on the anesthesiologists' experience and intuition. Recently, deep learning algorithms using invasive arterial pressure monitoring showed the good predictive ability of intraoperative hypotension. It can help the clinician's decisions. However, most patients undergoing general surgery are monitored by non-invasive parameters. Therefore, the investigators investigate the prediction model for intraoperative hypotension using non-invasive monitoring.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are included in the open database, VtialDB.
* The patients who underwent inhaled general anesthesia for non-cardiac surgery.
* The patients who have non-invasive monitoring data including blood pressure, electrocardiography, pulse oximetry, bispectral index, and capnography.

Exclusion Criteria:

* The patient with missing data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population included patients who underwent inhaled general anesthesia for non-cardiac surgery between June 2016 and August 2017 at Seoul National University Hospital, Seoul, South Korea.
Sampling Method: Probability Sample
Enrollment: 5175 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Deep learning model's prediction ability on intraoperative hypotension event | through study completion, an average of 3 hour
  Area under the curve the receiver operating characteristic (AUROC) curve for the deep learning model to predict intraoperative hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Lee HC, Chu YS, Song SW, Ahn GJ, Lee H, Yang S, Koh SB. Deep learning models for the prediction of intraoperative hypotension. Br J Anaesth. 2021 Apr;126(4):808-817. doi: 10.1016/j.bja.2020.12.035. Epub 2021 Feb 6. PMID 33558051
- [Background] Lee HC, Jung CW. Vital Recorder-a free research tool for automatic recording of high-resolution time-synchronised physiological data from multiple anaesthesia devices. Sci Rep. 2018 Jan 24;8(1):1527. doi: 10.1038/s41598-018-20062-4. PMID 29367620